CLINICAL TRIAL: NCT06980740
Title: Video-Tumorboard PLUS
Acronym: vTB+
Status: Recruiting | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); University Hospital, Bonn (Other); University Hospital Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: BO ff (Multi)-EK-16012025; 2025-275-b-S (Other: Ethikkommission Westfalen-Lippe)
Record Dates: First submitted 2025-04-16; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Malignant Melanoma; Telemedicine
Keywords: Malignant Melanoma; Telemedicine
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Retrospective
- 2: Prospective

SUMMARY:
In weekly expert meetings for oncological diagnostics and therapy, known as tumor boards, individual therapy recommendations are developed for cancer patients. By further developing and optimizing the CCCs' video tumor boards, initially using skin cancer as an example, we want to ensure that more patients can benefit from the expertise of several specialist disciplines and innovations - regardless of where they live.

ELIGIBILITY:
Inclusion Criteria:

* The study includes adult, external patients who, according to the certification requirements of the German Cancer Society, should be presented to the CCCs in a tumor board .

Inclusion criteria for patients:

* Minimum age 18 years
* Consent to participate in the study (signing of patient consent) should be presented in vTB+ according to the doctor, based on the disease/diagnosis, especially in the case of:

  * Malignant melanoma from stage IIB
  * Malignant melanoma and stage shift/recurrence o Extracutaneous melanoma o Cutaneous lymphoma from stage Ib o Problem cases with malignant, epithelial tumors (BCC, SCC) with interdisciplinary issues, e.g. complicated localization, extension/ infiltration (e.g. Ulcus rodens, Ulcus terebrans), metastasized tumors, immunosuppressed patients o all rare malignant skin tumors (including Merkel cell carcinoma, DFSP, MFH, leiomyosarcoma, S., Kaposi's sarcoma, angiosarcoma), regardless of stage o severe side effects from drug-based tumor therapy • is an external patient: An external patient is someone who receives tumor therapy exclusively or in co-treatment in the branch or in an external clinic (in distinction to patients without prior treatment for initial presentation at the CCC) . This also applies to patients who are only seen once at the vTB.

In this case, revenue/cost aspects and the DKG requirement are ignored. This means that so-called external patients can also be treated at the center, including initiation of therapy. The decisive factor is the presentation of the external patient (personal presentation of the external patients is not mandatory) and that external co-treaters are consistently informed and involved.

Inclusion criteria for external doctors:

* has a medical license
* has dermatological patients who are eligible to be presented in the vTB+

Exclusion Criteria:

Patients will be excluded from the study if they meet the following criteria:

* Linguistic or other limitations (such as dementia) that prevent independent consent to the privacy policy.
* No consent to participate in the study (patient consent) or withdrawal of consent during the course of the study In addition, external physicians will be excluded from the study if no joint cooperation agreement can be negotiated and signed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As part of the vTB+ study, an evaluation of the video tumor board is to be carried out for as broad a section of the population as possible. Women of childbearing potential with and without contraception make up a relevant proportion of the population. Participation in the study is not associated with physical interventions, so that the contraceptive status of fertile participants is irrelevant. Even in the case of pregnancy, participation in the study would be harmless. The exclusion of women of childbearing potential with and without contraception from the vTB+ study would therefore represent a gender-based disadvantage.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Presentation of external patients in the video-tumorboard | Day 365
  Increase in the proportion of external patients in the video-tumorboard

SECONDARY OUTCOMES:
Increase in the proportion of external patients invited to a clinical study | Day 365
  Increase in the proportion of external patients in clinical studies
Adherence to tumorboard recommendations for external patients | Up to two weeks after inclusion
  Proportion of implemented tumorboard recommendations for external patients
Offer of supportive therapies by the comprehensive cancer center | Up to two days after inclusion
  Proportion of (external) patients who are offered at least one supportive therapy (e.g. psychooncology) within the video-tumorboard
Duration of the transmission of the tumorboard recommendations | Up to two weeks after inclusion
  Duration of the transmission of the tumorboard recommendations
"Time to integration" into palliative care | Once per patient within two weeks after transmission of the tumorboard recommendation if applicable
  Time between medical recommendation for palliative care and first contact with palliative care

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Lenz, MD, Principal Investigator — Westdeutsches Tumorzentrum Münster, Universitätsklinikum Münster
Locations (3):
- Germany (3):
  - Abteilung für Integrierte Onkologie - CIO Bonn, Universitätsklinikum Bonn, Bonn
  - Nationales Centrum für Tumorerkrankungen Klinik u. Poliklinik für Dermatologie, Universitätsklinikum Dresden, Dresden
  - Westdeutsches Tumorzentrum Münster, Universitätsklinikum Münster, Münster

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol